CLINICAL TRIAL: NCT00030797
Title: A Randomized Phase II Trial Of Capecitabine And Different Schedules Of Irinotecan As First Line Treatment For Advanced Or Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/00; EU-20141
Record Dates: First submitted 2002-02-14; First posted 2003-06-25 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Irinotecan i.v. 70 mg/m2, day 1, 8, 15, 22, 29; Capecitabine p.o. 2 x 1000 mg/m2, d1-14, d22-35;
  Interventions: Drug: Irinotecan 70 mg/m2
- Arm B (Active Comparator): Irinotecan i.v. 240 mg/m2 day 1 and day 22; Capecitabine p.o. 2 x 1000 mg/m2, d1-14, d22-35;
  Interventions: Drug: Irinotecan 240 mg/m2

INTERVENTIONS:
Drug: Irinotecan 70 mg/m2 — Irinotecan i.v. 70 mg/m2, day 1, 8, 15, 22, 29
  Arms: Arm A
Drug: Irinotecan 240 mg/m2 — Irinotecan i.v. 240 mg/m2 day 1 and day 22
  Arms: Arm B

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combination chemotherapy in treating patients who have advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of different schedules of irinotecan in combination with capecitabine as first-line therapy, in terms of objective response rate, in patients with advanced or metastatic colorectal cancer.
* Compare the time to treatment failure, time to progression, and overall survival of patients treated with these regimens.
* Compare the safety profile, in terms of toxicity, of these regimens in these patients.
* Determine the quality of life in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (0 vs 1); disease symptoms, including pain, weight loss, loss of appetite, malaise, and fever of unknown origin (yes vs no); weight loss during the past 6 months (more than 5% vs 5% or less); and disease-free interval (more than 6 months vs 6 months or less). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive irinotecan IV over 1 hour on days 1, 8, 15, 22, and 29 and oral capecitabine twice daily on days 1-14 and 22-35.
* Arm II: Patients receive irinotecan IV over 1 hour on days 1 and 22 and oral capecitabine as in arm I.

Treatment in both arms repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on day 1 of each course, and at the first visit after treatment failure.

Patients are followed every 12 weeks for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 28-74 patients (14-37 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced or metastatic colorectal cancer

  * Unresectable disease
* At least 1 bidimensionally measurable lesion

  * At least 2 cm in perpendicular diameters
* No evidence of CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.25 times ULN

Cardiovascular:

* No clinically significant cardiac disease
* No congestive heart failure
* No New York Heart Association class III or IV heart disease
* No symptomatic coronary artery disease
* No uncontrolled cardiac arrhythmia
* No myocardial infarction within the past year

Gastrointestinal:

* No evidence of dysphagia
* No malabsorption or intestinal obstruction that would affect absorption or excretion of study drugs
* No chronic diarrhea

Other:

* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No psychiatric disability that would preclude study compliance
* No other significant medical condition
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for advanced or metastatic disease

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* At least 4 weeks since prior major surgery to the gastrointestinal tract

Other:

* No concurrent therapy for history of seizures or CNS disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2001-02; Primary Completion 2002-05 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus M. Borner, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern, Bern, Switzerland

REFERENCES:
- [Result] Borner MM, Bernhard J, Dietrich D, Popescu R, Wernli M, Saletti P, Rauch D, Herrmann R, Koeberle D, Honegger H, Brauchli P, Lanz D, Roth AD; Swiss Group for Clinical Cancer Research (SAKK), Berne, Switzerland. A randomized phase II trial of capecitabine and two different schedules of irinotecan in first-line treatment of metastatic colorectal cancer: efficacy, quality-of-life and toxicity. Ann Oncol. 2005 Feb;16(2):282-8. doi: 10.1093/annonc/mdi047. PMID 15668285